CLINICAL TRIAL: NCT00924521
Title: Grains Reduce Adiposity and Improve Nutrition Study (GRAINS) Increased Whole Grain Intake - Beneficial Effects on Visceral Adiposity, Vascular Function and Glucose Metabolism/Insulin Resistance
Brief Title: Grains Reduce Adiposity and Improve Nutrition Study
Acronym: GRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKE GRAIN
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome; Insulin Resistance
Keywords: grains; fiber; metabolic syndrome; insulin
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Refined grain (Active Comparator): Participants in this group will receive only refined grains as typically consumed in the average American diet.
  Interventions: Dietary Supplement: Refined grain
- Whole grain diet (Experimental): Participants in this group will receive 6-9 servings of whole grain daily to replace the refined grains typically included in the average American diet. Number of servings will depend upon calorie assignment.
  Interventions: Dietary Supplement: Whole grain diet

INTERVENTIONS:
Dietary Supplement: Whole grain diet — Participants in this group will receive 6-9 servings of whole grain daily to replace the refined grains typically included in the average American diet. Number of servings will depend upon calorie assignment.
  Arms: Whole grain diet
Dietary Supplement: Refined grain — Participants in this group will receive only refined grains as typically consumed in the average American diet.
  Arms: Refined grain

SUMMARY:
Whole grain intake beneficially affects body weight, body fat and glucose metabolism, and the investigators' previous work has shown that a high whole grain intake significantly reduced body fat in the abdominal region as measured by dual energy X-ray absorptiometry (DEXA) compared to a refined grain intake. Additional research is needed with regard to the mechanisms by which whole grains may affect visceral adiposity and the adipokines, which have been associated with risk for insulin resistance and type 2 diabetes. Therefore the proposed study aims to address these issues and in addition, includes exploratory work with adipocytes in cell culture to evaluate the effects of whole grains on adipocyte function.

Hypothesis:

There will be a greater reduction in visceral adiposity, indicators of insulin resistance (HOMA score), improvement in inflammatory status and improvement in adipokine levels after six weeks of a weight stable period and after six weeks of weight loss in subjects consuming 6-9 servings compared to 0 servings of whole grains per day.

DETAILED DESCRIPTION:
Including whole grains as part of a heart-healthy diet has been shown to be beneficial in decreasing body weight and body fat. The beneficial effects of whole grains on body weight may be explained by the larger volume and relatively low energy density of whole grain food thus leading to increased satiation. Reducing visceral fat is of particular importance as visceral adiposity has been associated with increased risk for metabolic diseases and cardiovascular disease.

The proposed study is a randomized, 2-parallel arm controlled feeding study. Subjects will be fed one of two weight maintenance diets (refined grain and whole grain) for 6 weeks, followed by a 6 week controlled weight loss period where subjects are fed the same diets, but at a reduced calorie level, designed to elicit weight loss (~2 lbs per week). Diets for both groups will have the same nutrient profile (percent of calories from fat, protein, carbohydrates, etc.); however, the whole grain (WG) group will substitute whole grains for refined grains in their grain intake (breads, tortillas, cereals, etc.). The WG group will be expected to take in 6-9 servings of whole grains per day on both diets. Plasma endpoints will be measured at baseline and at the end of the 6-week diet periods. Blood samples also will be taken at the mid-point of each period and held for analysis if deemed appropriate after initial data is reviewed. Endo-PAT will be conducted at baseline and at the end of each diet period as well as DEXA and MRI testing.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 to < 42
* Waist circumference of > 40 inches for males and > 35 inches for females and having one other of the criteria for metabolic syndrome will be recruited
* In this population, we will also accept the following:

  * LDL-C < 175 mg/dL
  * HDL-C > 25 mg/dL
  * Triglycerides < 400 mg/dL
* All subjects will be required to meet one specific criteria for metabolic syndrome beyond increased waist circumference

Exclusion Criteria:

* Smokers
* Have insulin-dependent diabetes
* Are pregnant or expecting to be pregnant, lactating in the last 6 months
* Are taking NSAIDS or other medications known to affect inflammatory markers or drugs affecting glucose metabolism

Blood pressure lowering medications are acceptable if the person has controlled BP at screening, <140/90 mmHg.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Body Composition | Week 6 and 12 - End of diet period 1 and 2
  To assess regional changes in body fat deposition, subjects will undergo a dual energy X-ray absorptiometry (DXA) scan at baseline (beginning of study) and end of each intervention period. Waist circumference measurements also will be taken at this time to track how much fat is lost from the abdominal area of the body.

SECONDARY OUTCOMES:
Fasting glucose | Time 0, week 6 and week 14 - Baseline end of each diet period
  Twelve-hour fasting blood samples (30ml) will be collected for analyses of plasma glucose levels.
Plasma cytokines | Week 0, week 6 and week 14 - Baseline end of each diet period
  Twelve-hour fasting blood samples (30ml) will be collected for analyses of plasma C-reactive protein and inflammatory cytokines. Blood samples obtained at baseline will be used to measure baseline values for study endpoints, whereas blood samples obtained at the end of each diet period will measure final endpoint values.
Endothelial Health | Week 0, week 6 and week 14 - Baseline end of each diet period
  Study subjects will undergo endothelial health assessment by EndoPAT analysis. The EndoPat procedure will occur while the subject is lying down in a relaxed state. Throughout the study, the inflation pressure of the EndoPAT device will be electronically set to 10mm Hg below diastolic BP. Testing begins with 10 min of rest. Following rest, baseline pulse amplitude is measured from each fingertip for 5 min. Next, arterial flow is interrupted for 5 min by a cuff placed on the forearm at an occlusion pressure of 250 mmHg. Following occlusion release, pulse amplitude recording continues for 5 min.
Resting Metabolic Rate | Week 0 and week 14 - Baseline and end of diet period 2
  The COSMED Fitmate is a state-of-the-art resting metabolic rate machine that takes accurate, quick readings of your oxygen use. Participants will lie quietly without moving for 30 minutes upon arrival. A mask will be placed around the nose and mouth and participant will be asked to remain still for another 15 min will resting metabolic rate is measured. The test provides valuable information about how much energy (calories) an individual burns in a 24-hour period. The test will take ~15 min to complete.
Appetite Hormones | Week 0, week 6 and week 14 - Baseline end of each diet period
  Twelve-hour fasting blood samples (30ml) will be collected to assess changes in plasma appetite hormones across the two diet periods.
Abdominal obesity | Week 14 - End of diet period 2
  A subset of subjects will undergo magnetic resonance imaging (MRI) scans in the abdominal region by standard protocols. Subjects will be placed in a prone position in the magnet with their arms stretched above their head. A series of 40-47 T1-weighed axial spin echo images, will be taken in the abdominal region using established body landmarks. Body compartment volumes for total abdominal and visceral adipose tissue, as well as muscle, will then be obtained by tissue integration analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Result] Katcher HI, Legro RS, Kunselman AR, Gillies PJ, Demers LM, Bagshaw DM, Kris-Etherton PM. The effects of a whole grain-enriched hypocaloric diet on cardiovascular disease risk factors in men and women with metabolic syndrome. Am J Clin Nutr. 2008 Jan;87(1):79-90. doi: 10.1093/ajcn/87.1.79. PMID 18175740
- [Derived] Harris Jackson K, West SG, Vanden Heuvel JP, Jonnalagadda SS, Ross AB, Hill AM, Grieger JA, Lemieux SK, Kris-Etherton PM. Effects of whole and refined grains in a weight-loss diet on markers of metabolic syndrome in individuals with increased waist circumference: a randomized controlled-feeding trial. Am J Clin Nutr. 2014 Aug;100(2):577-86. doi: 10.3945/ajcn.113.078048. Epub 2014 Jun 18. PMID 24944054